CLINICAL TRIAL: NCT04909242
Title: A Phase 1 Randomised, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of DZD9008 Following Single Ascending Dose and the Effect of Low-fat Meal on Pharmacokinetics of DZD9008 in Healthy Adult Participants
Brief Title: Assessing the Safety, Tolerability and Pharmacokinetics(PK) of DZD9008 and the Effect of Low-fat Meal on PK of DZD9008 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DZ2021E0004
Record Dates: First submitted 2021-05-13; First posted 2021-06-01 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- single oral dose of DZD9008 (Experimental): single dose of DZD9008 (50 mg, 100 mg, 200 mg, 300 mg and 400 mg, tablet)
  Interventions: Drug: DZD9008
- single oral dose of placebo (Placebo Comparator): single dose of placebo (matching placebo, 50 mg, 100 mg, 200 mg, 300 mg and 400 mg, tablet)
  Interventions: Drug: Placebo
- single oral dose of DZD9008 (300 mg, tablet) (Experimental)
  Interventions: Drug: DZD9008
- single oral dose of DZD9008 (100 mg, tablet or suspension) (Experimental)
  Interventions: Drug: DZD9008

INTERVENTIONS:
Drug: DZD9008 — In the double blind, randomised, placebo-controlled trial (Part A - SAD), healthy adult participants will be randomized to receive DZD9008 at different dose levels. There are 5 planned dose cohorts, starting from 50 mg once daily. If tolerated, subsequent cohorts will test increasing doses of DZD9008 or matching placebo, namely 100 mg, 200 mg, 300 mg and 400 mg.
  Arms: single oral dose of DZD9008
Drug: Placebo — In the double blind, randomised, placebo-controlled trial (Part A - SAD), healthy adult participants will be randomized to receive matching placebo for DZD9008 at different dose levels. There are 5 planned dose cohorts of matching placebo for DZD9008, starting from 50 mg once daily.
  Arms: single oral dose of placebo
Drug: DZD9008 — In Part C, healthy adult participants will be enrolled to receive a single dose of DZD9008 as suspension in period 1 and as tablet in period 2.
  Arms: single oral dose of DZD9008 (100 mg, tablet or suspension)
Drug: DZD9008 — Healthy adult participants will be randomized to receive DZD9008 single dose at a defined dose under a cross-over condition with or without food (low-fat in Part B; high-fat in Part D).
  Arms: single oral dose of DZD9008 (300 mg, tablet)

SUMMARY:
This is a Phase 1, randomised, double-blind, placebo-controlled, single ascending dose sequential group study in healthy participants. This study consists of three parts: Part A (single dose escalation, SAD) , Part B (food effect, FE) and Part C (relative bioavailability, BA).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand the nature of the trial and provide a signed and dated, written informed consent form before any study-specific procedures, sampling and analyses.
* Provision of signed and dated written Optional Genetic Research informed consent prior to collection of samples for optional genetic research.
* Healthy male or female participants aged 18 to 60 years (inclusive), with BMI 18.0 to 30.0 kg/m2 (inclusive). Body weight: ≥ 55 kg for male, ≥ 45 kg for female.
* Healthy participants defined as the absence of acute or chronic clinically significant deviations from normal in medical history, physical examination, visual assessment, electrocardiogram (ECG), and clinical laboratory determinations at screening.
* Participants must agree to practice effective contraception.
* Normal baseline PFTs (≥ 80% predicted normal for spirometry, lung volumes).
* Normal baseline ECG (QTcF < 450 msec, PR < 210 msec).
* Non-smoker (not smoked within 3 months).
* Liver biochemistry parameters: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN); Total bilirubin ≤ 1.5 × ULN
* Adequate organ function including hepatic, renal, cardiac, visual and bone marrow function as determined by the investigator.

Exclusion Criteria:

* Ongoing or prior pulmonary disease including asthma, chronic obstructive pulmonary disease, interstitial lung disease and pneumonitis including but not limited to drug-related pneumonitis.
* Women who are breast feeding.
* Positive pregnancy test prior to study entry.
* History of malignancy of any type, with the exception of the following: surgically excised non-melanomatous skin cancers more than 5 years prior to receiving IP.
* A history of additional risk factors for TdP (e.g. heart failure, hypokalemia, family history of Long QT syndrome).
* No prior history of atrial fibrillation within 6 months prior to first dosing of DZD9008
* Manifestations of malabsorption due to prior GI surgery, GI disease, or for an unknown other reason that may affect the absorption of DZD9008-. Pulmonary infections or other active infection within 30 days of informed consent
* History of bleeding disorder (including hemophilia, Von Willebrand disease, etc), history of stroke or intracranial haemorrhage within 6 months before study drug administration.
* Judgement by the investigator that the participant is not likely to comply with study procedures, restrictions and requirements.
* Positive serology or a known history of hepatitis B virus (HBV), hepatitis C virus (HCV), HIV.
* Resting blood pressure > 140/90 mmHg at screening .
* Resting pulse rate < 45 beats per minute.
* History of severe allergy or hypersensitivity reaction or ongoing allergy or hypersensitivity reaction, as judged by investigator, or history of hypersensitivity to EGFR/HER2/BTK inhibitors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 14 days after study drug administration
  To assess the safety and tolerability of DZD9008 following oral administration of single ascending doses in healthy adult participants.
Number of participants with clinically significant laboratory assessment abnormalities | up to 14 days after study drug administration
  To assess the safety and tolerability of DZD9008 following oral administration of single ascending doses in healthy adult participants.
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | up to 14 days after study drug administration
  To assess the safety and tolerability of DZD9008 following oral administration of single ascending doses in healthy adult participants.
Number of participants with clinically significant abnormalities in LVEF | up to 14 days after study drug administration
  To assess the safety and tolerability of DZD9008 following oral administration of single ascending doses in healthy adult participants.
Number of participants with clinically significant abnormalities in FEV1% | up to 14 days after study drug administration
  To assess the safety and tolerability of DZD9008 following oral administration of single ascending doses in healthy adult participants.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of DZD9008 | up to 10 days after study drug administration
Time to reach maximum plasma concentration (tmax) | up to 10 days after study drug administration
Area under the concentration-time curve from time 0 (pre-dose) to the time of the dosing interval (AUC0-t) | up to 10 days after study drug administration
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | up to 10 days after study drug administration
Apparent total plasma clearance (CL/F) | up to 10 days after study drug administration
Apparent volume of distribution (Vz/F) | up to 10 days after study drug administration
Mean residence time (MRT) | up to 10 days after study drug administration
Terminal elimination half-life (t1/2) | up to 10 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No